CLINICAL TRIAL: NCT00891852
Title: Non-Invasive Determination of Fetal Chromosome Abnormalities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lenetix Medical Screening Laboratory (Industry)
Responsible Party: Leonard Kellner, Lenetix, Inc.
Other Study IDs: 110106-1
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Down Syndrome (Trisomy 21); Edward's Syndrome (Trisomy 18); Patau Syndrome (Trisomy 13); Klinefelter Syndrome (47, XXY); and Other Chromosome; Abnormalities.
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome; Klinefelter Syndrome; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The overall significance of this study is to develop a laboratory developed test (LDT) to use a new marker in the maternal blood to better identify pregnancies that have a child with a chromosome abnormality such as Down syndrome (trisomy 21), Edward's syndrome (trisomy 18), Patau syndrome (trisomy 13), Klinefelter syndrome, (47, XXY), and other chromosome abnormalities. Accomplishing that task would reduce the need for invasive amniocentesis and CVS procedures.

ELIGIBILITY:
Inclusion Criteria:

* This study is only applicable to women who are between 8 and 30 weeks' gestation and who have been determined increased risk for fetal aneuploidy. In the interest of expediting and simplifying this study, the investigators want only women who have already decided to undergo second-trimester amniocentesis or CVS.

Exclusion Criteria:

* The only exclusion criteria are those mentioned.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators anticipate enrolling 1000 subjects who are presenting for prenatal diagnosis by CVS or genetic amniocentesis for increased risk for fetal aneuploidy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Brown, MD, Principal Investigator — Lenetix, Inc.
Locations (7):
- United States (7):
  - Maryland Perinatal Associates, Rockville, Maryland
  - Atlantic Maternal Fetal Medicine, Moristown, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Elite Women's Health, New Hyde Park, New York
  - Columbia University, NewYork-Presbyterian Hospital, New York, New York
  - New York Perinatal Associates, New York, New York
  - UVM, Burlington, Vermont